CLINICAL TRIAL: NCT00323258
Title: PILOT-EBM: Patient Focused Intervention to Improve Long-term Adherence to Evidence Based Medications
Brief Title: Study of an Intervention to Improve Use of Life-saving Medications for Heart Disease
Acronym: PILOT-EBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Pro00005018; U18HS010548 (AHRQ)
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-05

CONDITIONS: Cardiovascular Disease
Keywords: Heart disease; Coronary disease; Patient compliance; Treatment refusal; Pharmacists; Continuity of patient care; Evidence-based medicine; Patient education; Adherence
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Patient Compliance; Treatment Refusal | interventions — Educational Status; Pharmacists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients enrolled in the intervention arm received inpatient education on the importance of medication and assessment of barriers to adherence. A pill box, pocket medication card, and tips for remembering to take medications were provided. The community pharmacist was notified of the subject's enrollment. The community pharmacist was asked to reinforce importance of evidence-based medications and assess the subject's medication adherence every 6 weeks for 6 months. If a problem was noted, the subject's health care team will be notified.
  Interventions: Behavioral: oral education & written tips for remembering medications; Device: pill box; Device: pocket medication card; Behavioral: sharing information with community pharmacist; Behavioral: Medication use evaluations by community pharmacist; Behavioral: informing physician if patient has stopped a medication; Behavioral: Routine discharge counseling; Other: Letter to physician/discharge summary
- Usual Care (Active Comparator): The usual care group received routine discharge counseling performed by the patient-care nurse and a letter/discharge summary from the hospital physician to the community physician listing the discharge medications, procedures, and recommendations. Enrolled patients in the usual care arm were not disclosed to the community pharmacy until the end of the study period when refill records were requested.
  Interventions: Behavioral: Routine discharge counseling; Other: Letter to physician/discharge summary

INTERVENTIONS:
Behavioral: oral education & written tips for remembering medications — Clinical pharmacist will review purpose of medications of interest (beta-blockers, statins, Angiotensin Converting Enzyme Inhibitor (ACEI)/Angiotensin Receptor Blocker (ARB), aspirin, and other anti-platelets) with the subject. A written list of tips for remembering medications will be provided and reviewed.
  Other Names: Cue-dose training
  Arms: Intervention
Device: pill box — Subject is provided a pill box and briefly instructed on how to use the box.
  Other Names: Pill box organizer; pillbox
  Arms: Intervention
Device: pocket medication card — Subject is provided with a card that contains space for prescription and non-prescription medications. If desired the clinical pharmacist-investigator will complete the card for the subject.
  Other Names: Medication List; List of Medications
  Arms: Intervention
Behavioral: sharing information with community pharmacist — A fax is sent to the designated community pharmacy at the time of the subject's discharge from the hospital. The fax contains the subject's medications of interest, barriers to medication adherence, and physicians' contact information.
  Other Names: increased communication with community pharmacist
  Arms: Intervention
Behavioral: Medication use evaluations by community pharmacist — The community pharmacist will assess use of medications of interest at time of first medication fill and by reviewing the subject's computerized medication profile at the pharmacy. Assessments occur at first visit to pharmacy, 6-weeks, 12-weeks, 18-weeks, and 24-weeks. If there are issues with any medications of interest the subject will be called. If needed, the subject's health care team will be notified.
  Other Names: medcation adherence verification
  Arms: Intervention
Behavioral: informing physician if patient has stopped a medication — The community pharmacist or clinical pharmacist-investigator will fax the subject's physician to notify that a medication has been stopped.
  Other Names: Communication with physician about patient's medication use
  Arms: Intervention
Behavioral: Routine discharge counseling — Both groups received routine discharge counseling performed by the patient-care nurse.
  Other Names: Discharge instructions
Other: Letter to physician/discharge summary — A letter/discharge summary from the hospital physician to the community physician listing the discharge medications, procedures, and recommendations.
  Other Names: Communication to physician about hospital course.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a program to help patients with heart disease stay on their heart medications.

DETAILED DESCRIPTION:
Heart disease is the leading cause of death for men and women in the United States. For patients with documented coronary artery disease (CAD), anti-platelet agents, beta-blockers and statins have all been shown to improve survival and reduce the frequency of myocardial infarction. Yet, previous research by the Duke CERTs has shown that in a population of over 28,000 patients with documented CAD, only 21% reported consistent use of triple therapy with aspirin, beta-blockers and lipid lowering therapy. These results stimulated the Duke CERTs to devise an intervention to improve adherence to these life-saving medications.

Comparisons: Patients admitted to Duke University Hospital or Southeastern Regional Medical Center (SRMC) with CAD or CAD plus heart failure who agree to participate, will be randomized to an intervention or control arm. The control group will receive usual care, which consists of routine discharge counseling performed by the patient-care nurse and a letter/discharge summary from the Duke physician to the community physician. In addition to usual care, the intervention group will receive focused medication counseling in the hospital by the clinical pharmacist-investigator, who will identify and address potential barriers to medication adherence and will reinforce the importance of taking evidence-based medications long term. Discharge medications will be shared with the community pharmacist. The community pharmacist will monitor for problems with adherence and communicate issues back to the patient and the patient's care team.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Utilize a pharmacy in Durham, Robeson, Person, Granville, or Vance County, NC
* Have coronary artery disease (CAD) documented in the medical record by one of the following:

  1. A diagnosis of unstable angina or acute myocardial infarction (ST segment elevation or non-ST segment elevation myocardial infarction)
  2. A cardiac catheterization demonstrating CAD greater than or equal to 50 narrowing of artery)
  3. Prior angioplasty
  4. Prior coronary artery stent
  5. Prior coronary artery bypass graft surgery (CABG)
* Plan to have their prescription medications filled and refilled by one of the participating pharmacies
* Prescribed aspirin or another antiplatelet, a beta-blocker and statin agent (referred to as triple therapy for this study) at discharge. If a patient has a true contraindication to any of the three medication groups in triple therapy, they will still be eligible for the study

Exclusion Criteria:

* Providers predict an anticipated hospital stay of less than 48 hours
* Patient plans to use a pharmacy outside of Durham, Robeson, Person, Granville, or Vance County, NC
* Patient is unable to give consent (cognitively impaired, does not speak English, or has altered mental status)
* Patient transferred to Cardiothoracic Surgery service for CABG
* Patient has terminal condition and may not survive until 6-month follow-up
* Patient lives in a correctional or long-term care facility
* Patient will be unable to participate in follow-up phone call (hearing impaired without caregiver who can help or does not have a phone)
* Patient is a known participant in the Duke Heart Failure Program
* Patient does not agree to use only the one Durham, Robeson, Person, Granville, or Vance County pharmacy throughout the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2006-06; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith M. Kramer, MD,MS, Principal Investigator — Duke University; Nancy Allen LaPointe, PharmD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Newby LK, LaPointe NM, Chen AY, Kramer JM, Hammill BG, DeLong ER, Muhlbaier LH, Califf RM. Long-term adherence to evidence-based secondary prevention therapies in coronary artery disease. Circulation. 2006 Jan 17;113(2):203-12. doi: 10.1161/CIRCULATIONAHA.105.505636. Epub 2006 Jan 9. PMID 16401776
- [Result] Calvert SB, Kramer JM, Anstrom KJ, Kaltenbach LA, Stafford JA, Allen LaPointe NM. Patient-focused intervention to improve long-term adherence to evidence-based medications: a randomized trial. Am Heart J. 2012 Apr;163(4):657-65.e1. doi: 10.1016/j.ahj.2012.01.019. PMID 22520532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients hospitalized at Duke University Hospital (Durham, NC) were screened for study enrollment from July 5, 2006, through July 2, 2009. To increase enrollment, the study was opened to enrollment at Southeastern Regional Medical Center (Lumberton, NC) on May 27, 2008.
Pre-assignment Details: After patients provided written informed consent, the study pharmacist collected baseline demographics, medical history, medication history, potential barriers to medication adherence, pharmacy name, physicians' contact information, and the Beliefs about Medicines Questionnaire (BMQ).
Groups:
- Intervention Arm: Patients enrolled in the intervention arm received inpatient education on the importance of medication and assessment of barriers to adherence. A pill box, pocket medication card, and tips for remembering to take medications were provided. The community pharmacist was notified of the subject's enrollment. The community pharmacist was asked to reinforce importance of evidence-based medications and assess the subject's medication adherence every 6 weeks for 6 months. If a problem was noted, the subject's health care team will be notified.
  The intervention arm originally contained 71 subjects, 55 completed the 6 month follow-up phone call and 57 had refill records available at 6 months post-discharge. The periods listed here represent the same 6 month period with different numbers of particpants having the phone call or refill records available.
- Usual Care: The usual care group received routine discharge counseling performed by the patient-care nurse and a letter/discharge summary from the hospital physician to the community physician listing the discharge medications, procedures, and recommendations. Enrolled patients in the usual care arm were not disclosed to the community pharmacy until the end of the study period when refill records were requested.
  The control arm originally contained 72 subjects, 53 completed the 6 month follow-up phone call and 58 had refill records available at 6 months post-discharge. The periods listed here represent the same 6 month period with different numbers of particpants having the phone call or refill records available.
Period: Primary Outcome (Phone Call at 6 Months)
Arm/Group | Intervention Arm | Usual Care
Started | 71 | 72
Completed | 55 | 53
Not Completed | 16 | 19
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 12 | 11
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Died between 180-240 days (call period) | 2 | 1
Period: Secondary Outcome (6 Mon Refill Records)
Arm/Group | Intervention Arm | Usual Care
Started | 71 | 72
Completed | 57 | 58
Not Completed | 14 | 14
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 12 | 10
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Usual Care | Total
Number analyzed (Participants) | 71 | 72 | 143
Age Continuous [Median (Inter-Quartile Range); unit: years] | 63 [54 to 71] | 62 [52 to 70] | 62 [53 to 70]
Age Continuous [Mean (Standard Deviation); unit: years] | 63.0 (11.5) | 61.5 (12.0) | 62.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 47 | 44 | 91

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Adherence to Triple Therapy (Aspirin/Antiplatelet; Beta Blocker; and Statin) at 6 Months
Description: Percent of patients in each group adherent to triple therapy (aspirin/antiplatelet; beta blocker; and statin) 6 months after discharge as assessed by medication history obtained during a follow-up phone call by a blinded pharmacist
Time Frame: 6 months
Population: Those participants alive and able to speak to pharmacist on 6 month follow up phone call. Missing (n=35)- Could not be reached: 12 intervention and 11 usual care, Died between 0-6 months: 1 intervention and 2 usual care, Died during call period: 2 intervention and 1 usual care, refused to participate in call: 1 intervention and 5 usual care.
Measure: Number; unit: percentage of participants
Groups:
- Intervention: Inpatient education on the importance of medication and assessment of barriers to adherence, pill box, pocket medication card, and tips for remembering to take medications. Community pharmacist reinforced importance of medications and assessed medication adherence every 6 weeks for 6 months. If a problem was noted, the subject's health care team will be notified.
- Usual Care: Routine discharge counseling performed by the patient-care nurse and a letter/discharge summary from the hospital physician to the community physician listing the discharge medications, procedures, and recommendations. Enrolled patients in the usual care arm were not disclosed to the community pharmacy until the end of the study period when refill records were requested.
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 55 | 53
percentage of participants | 91 | 94
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Sample size of 286 patients(143 patients per group).Based on an estimated absolute improvement in medication adherence of 15% in the intervention group (eg, 85% in the intervention group, 70% in the control group), a 2-sided test with α level of .05, a 15% dropout rate, and power of 0.80; Test type: Non-Inferiority or Equivalence — Equivalence analysis. Null hypothesis: The will be no difference in proportion of participants adherent to triple therapy in the "treatment" arm compared to those who receive "usual care."; p = .50, Chi-squared

2. Secondary Outcome: Percent of Patients Adherent to Beta-blocker and Statin Via Refill Records
Description: Percent of patients in each group adherent to beta-blocker and statin for 6 months after discharge as assessed by refill records from the patient's pharmacy
Time Frame: 6 months
Population: Those participants who were living, did not withdraw, and refill records were available from their pharmacy. Missing (n=28)- Refill records not available: 12 intervention and 10 usual care, Died between 0-6 months: 1 intervention and 2 usual care, Withdrew: 1 intervention and 2 usual care.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 57 | 58
percentage of participants | 53 | 38
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Sample Size calculated as 286 total or 143 patient per treatment group. Based on a baseline adherence rate of 70%, an estimated absolute improvement in medication adherence of 15.0% in the intervention group, we would require 122 patients per group assuming a 2-sided test with alpha-level of .05 and power of .80. To sustain a 15% dropout/ loss to follow-up rate, about 143 patients per group (286 patients total) would need to be consented; Test type: Non-Inferiority or Equivalence — Equivalence analysis. Null hypothesis: The will be no difference in the proportion of participants who are >/= 75% adherent to combined beta-blocker and statin therapy in the "treatment" arm compared to those who receive "usual care."; p = 0.11, Chi-squared

3. Secondary Outcome: Percent of Patients Adherent to Beta-blocker Via Refill Records
Description: According to the local pharmacy records, the patient has had a supply of beta-blocker for at least 75% of the days from the day of discharge to 180 days after the discharge date. Refill records from 90 days prior to index admission will be taken into account.
  % adherence = (days of available drug supply in the first 180 days/180)*100 If % adherence = or > 75, then adherence = yes
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of patients with PDC >or=75%
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 57 | 58
percentage of patients with PDC >or=75% | 71 | 49
Statistical Analysis 1: Comparison: Intervention vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Equivalence analysis. Null hypothesis: The will be no difference in the proportion of participants who are >/= 75% adherent to beta-blockers in the "treatment" arm compared to those who receive "usual care."; p = 0.03, Chi-squared

4. Secondary Outcome: Percent of Patients Adherent to Statin Via Refill Records
Description: According to the local pharmacy records, the patient has had a supply of statin for at least 75% of the days from the day of discharge to 180 days after the discharge date. Refill records from 90 days prior to index admission will be taken into account.
  % adherence = (days of available drug supply in the first 180 days/180)*100 If % adherence = or > 75, then adherence = yes
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of patients with >or=75%
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 57 | 58
percentage of patients with >or=75% | 58 | 49
Statistical Analysis 1: Comparison: Intervention vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Equivalence analysis. Null hypothesis: The will be no difference in the proportion of participants who are >/= 75% adherent to statins in the "treatment" arm compared to those who receive "usual care."; p = 0.34, Chi-squared

5. Secondary Outcome: Death in Intervention Patients Compared to Usual Care
Description: Number of patients who died in each treatment group prior to the 6 month follow-up time point.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 71 | 72
participants | 1 | 2

ADVERSE EVENTS:
Description: This was a behavioral and educational intervention. It was minimal risk and all patients (both groups) were taking the same medication classes. Adverse Events were not collected for this study. Death was not considered an event but collected only as a reason for not being available for follow-up with a participant.
Arm/Group | Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No